CLINICAL TRIAL: NCT07288021
Title: Topical Anesthesia During Catheter Insertion for Cervical Ripening (TOLERANCE)
Acronym: TOLERANCE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0061-23-BNZ
Record Dates: First submitted 2025-10-26; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Labor, Induced
Keywords: induction; balloon catheter; EMLA; Lidocaine/prilocaine; pain
MeSH Terms: conditions — Pain | interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both creams (EMLA and placebo) are specially made in similar containers, labeled as A and B. Head of pharmacy in the study's medical center alone is aware which is EMLA or placebo. Both substances are of similar smell, texture and color.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EMLA (Experimental)
  Interventions: Drug: Topical Analgesia with Lidocaine-Prilocaine cream
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topical Analgesia with Lidocaine-Prilocaine cream — patients allocated to 'EMLA' arm will receive topical analgesia cream prior to speculum insertion, as part of the administration of balloon catheter insertion process.
  3 puffs of the cream will be applied to the perineum, posterior fourchette and posterior vaginal wall by administrating physician. A pause of 7 minutes in the process will be made to allow for maximal analgesic affect.
  Arms: EMLA
Other: Placebo — patients allocated to 'Placebo' arm will receive lubrication with placebo cream prior to speculum insertion, as part of the administration of balloon catheter insertion process.
  3 puffs of the cream will be applied to the perineum, posterior fourchette and posterior vaginal wall by administrating physician. A pause of 7 minutes in the process will be made.
  Arms: Placebo

SUMMARY:
The goal of this RCT is to learn if application of topical anesthetic cream to the perineum and posterior wall of vagina prior to balloon catheter insertion as part of labor induction will reduce pain levels experienced by pregnant individuals.

All participants are 18 or older, carrying a singleton in vertex position and in need of labor induction, are late-preterm or term (34 weeks gestation and onward) and without contraindication to vaginal delivery.

Investigators seek to compare pain levels and patient satisfaction between two groups:

Nulliparous patients, using EMLA or placebo (randomized, double blinded). Multiparous patients, EMLA or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for labor induction with balloon catheter.
* 18 years of age or older.
* Singleton pregnancy with a cephalic presentation.
* ≥ 34 completed gestational weeks.
* Does not participate in any other trial that might affect maternal or fetal/neonatal outcomes.
* No contraindication for vaginal delivery

Exclusion Criteria:

* Unable or unwilling to provide and sign informed consent forms.
* Known sensitivity to EMLA or placebo substance.
* Known vulvodynia or vaginismus - rendering vaginal examination not possible.
* Any chronic pain syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain levels during insertion | directly after application and insertion of balloon catheter.
  Pain levels during insertion of balloon catheter, as experienced by participant and ranked from 1 to 5 [1 - no pain at all 2 - mild discomfort 3 -strong pain yet bearable 4 -severe pain 5 - unbearable pain (requires cessation of insertion)].

SECONDARY OUTCOMES:
analgesia while with balloon catheter | 6-12 hours
  need for medical analgetics while with balloon catheter, to be checked by analgetics given by nursing staff while the patient is with the balloon cathether in place - a dichotomic variable (yes/no).
pain score during removal of catheter | to be asked directly after removal, on a scale of 1-5.
  Pain levels during removal of balloon catheter, as experienced by participant and ranked from 1 to 5 [1 - no pain at all 2 - mild discomfort 3 -strong pain yet bearable 4 -severe pain 5 - unbearable pain (requires cessation of insertion)].
willingness to undergo cervical ripening with balloon catheter in the future | to be asked directly after removal, on a scale of 1-5.
  willingness to undergo cervical ripening with balloon catheter in the future, on a scale of 1-5 (1- no, not under any circumstances; 2 - only if no other option exists; 3 - ambivalent; 4 - yes, but with concern; 5 - yes, no problem).
analgesia during delivery | From time of balloon insertion until the time of delivery, assessed up to 3 days and to be checked immediately after delivery.
  need and use for medical analgetics during the delivery process, including epidural, dolestion and NO.
mode of delivery | at delivery
  mode of delivery - vaginal, operative vaginal of cesarean delivery
neonatal weight | immediately after delivery
  neonatal weight in grams and percentile according to birth weight curves
APGAR [Appearance (color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), and Respiration (breathing)] score | up to 10 minutes after delivery
  APGAR scores at 1, 5 and 10 minutes of life of newborn, as given by midwife/doctor present at the time. higher values on this score reflect a better outcome.
cord blood gas | up to 10 minutes after delivery
  cord blood gas levels, the first measurement taken after birth and up to 10 minutes after delivery.
Neonatal Intensive Care Unit (NICU) admission | from delivery and up to 1 week
  NICU admission of newborn within first week of life
neonatal infection | 1st week after delivery
  neonatal infection or suspicion of during birth hospitalization
duration of insertion procedure | balloon insertion duration, estimated as up to 20 minutes
  duration of insertion of catheter procedure
difficulty of insertion | to be reported by inserting doctor immediately after insertion procedure is completed, estimated up to 20 minutes.
  difficulty of insertion of catheter, as described by inserting physician
obstetric trauma | up to an hour after delivery
  presence of, and degree, of perineal lacerations

OTHER OUTCOMES:
Participant Satisfaction After Balloon Catheter Insertion | the patient is to be asked by inserting physician directly after insertion, on a scale of 1-5.
  satisfaction of participant from insertion of balloon catheter, as ranked by participant on a scale of 1-5 (1 - completely unhappy; 2 - slightly unhappy; 3 - ambivalent; 4 - mildly pleased; 5 - very pleased).

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided